CLINICAL TRIAL: NCT00643786
Title: Validation of a Kalinox's Administration Protocol for Dental Cares : Interest of Re-oxygenation and Pollution Control
Brief Title: Interest of Re-oxygenation After Inhalation of 50% Nitrous Oxide / 50% Oxygen Premix in Dental Cares
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Peter ONODY, MD, Air Liquide Santé International
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT : 031003
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Dental Cares Under Kalinox's Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Oxygène
  Interventions: Drug: Oxygène
- B (Placebo Comparator): Air Médical
  Interventions: Drug: Air Médical

INTERVENTIONS:
Drug: Oxygène — Flow of gas administrated to the patient between 4 and 15 litre/min during 5 minutes after the end of Kalinox's inhalation
  Arms: A
Drug: Air Médical — Flow of gas administrated to the patient between 4 and 15 litre/min during 5 minutes after the end of Kalinox's inhalation
  Arms: B

SUMMARY:
The usefulness of re-oxygenation after inhalation of 50% nitrous oxide and 50% oxygen premix (Kalinox 170 bar) during dental care is studied and the pollution resulting from administration of Kalinox is also investigated.

ELIGIBILITY:
Inclusion Criteria:

* From 1 year old
* anxious or phobic patients
* very young children requiring selective dental cares
* mental deficient patients
* ASA 1 or ASA 2 patients

Exclusion Criteria:

* ASA 3 or ASA 4 patients
* contraindication linked to the experimental product
* patients with mental disorder incompatible with the motory test
* patients that have received anxiolytic treatment less than 2 hours before the dental care

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2004-02; Primary Completion 2007-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Measurement of SpO2 | In continuous

SECONDARY OUTCOMES:
Analysis of ambient air pollution by nitrous oxide and patient's acceptance | In continuous

CONTACTS AND LOCATIONS:
Locations (1):
- UFR Odontologie Equipe d'accueil 3847, Clermont-Ferrand, France